CLINICAL TRIAL: NCT00006314
Title: Cytomegalovirus Spread and Reactivation in Blood Cells
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 922; R01HL063470 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2006-01

CONDITIONS: Blood Disease; Cytomegalovirus Infections
MeSH Terms: conditions — Hematologic Diseases; Cytomegalovirus Infections

SUMMARY:
To investigate the relationship between HCMV and bone marrow progenitor cells to understand whether HCMV is latent in CD34 + bone marrow progenitors and the mechanism by which the virus remains in a latent state.

DETAILED DESCRIPTION:
BACKGROUND:

Despite progress in understanding the pathophysiology of human cytomegalovirus (HCMV) infections, its manifestations in the immune compromised host are frequently associated with high morbidity and mortality. In this setting, HCMV disease can develop e.g. following immune suppression as a result of reactivation of latent HCMV acquired earlier in life. The mechanisms leading to establishment of latent infections and their subsequent reactivation are not clear. It is also unknown whether HCMV exists in a latent form with limited viral gene expression or as a persistent infection with normal virus transcription.

DESIGN NARRATIVE:

The specific aims of the study were to: 1) examine the percentage of HCMV positive donors whose bone marrow progenitors contained HCMV DNA using nested PCR and determine if virus could be rescued from those cells. 2) Analyze the HCMV life cycle in hematopoietic progenitor and stem cells. 3) identify and analyze HCMV gene expression in in vivo infected leukocytes. Bone marrow progenitors containing HCMV DNA detectable by nested PCR were isolated from human donors and used as as source of mRNA to prepare Cdna libraries. 4) Determine if gene(s) expressed in bone marrow progenitors were important in either establishing or maintaining a latent infection or in the lytic cycle of HCMV. Information provided from the above studies yielded information important in planning future approaches for the therapy of HCMV infections.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen St. Jeor — University of Nevada, Las Vegas

REFERENCES:
- [Background] Crapnell K, Zanjani ED, Chaudhuri A, Ascensao JL, St Jeor S, Maciejewski JP. In vitro infection of megakaryocytes and their precursors by human cytomegalovirus. Blood. 2000 Jan 15;95(2):487-93. PMID 10627453
- [Background] Rizvanov AA, van Geelen AG, Morzunov S, Otteson EW, Bohlman C, Pari GS, St Jeor SC. Generation of a recombinant cytomegalovirus for expression of a hantavirus glycoprotein. J Virol. 2003 Nov;77(22):12203-10. doi: 10.1128/jvi.77.22.12203-12210.2003. PMID 14581557
- [Background] Khaiboullina SF, Maciejewski JP, Crapnell K, Spallone PA, Dean Stock A, Pari GS, Zanjani ED, Jeor SS. Human cytomegalovirus persists in myeloid progenitors and is passed to the myeloid progeny in a latent form. Br J Haematol. 2004 Aug;126(3):410-7. doi: 10.1111/j.1365-2141.2004.05056.x. PMID 15257715
- [Background] Bego M, Maciejewski J, Khaiboullina S, Pari G, St Jeor S. Characterization of an antisense transcript spanning the UL81-82 locus of human cytomegalovirus. J Virol. 2005 Sep;79(17):11022-34. doi: 10.1128/JVI.79.17.11022-11034.2005. PMID 16103153